CLINICAL TRIAL: NCT03508024
Title: Patients With Alzheimer's Disease or Related Youth Disease
Acronym: PARMAAJJ
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: NI_2016_39; 2017-A00486-47 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-11-08; First posted 2018-04-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2018-04

CONDITIONS: Alzheimer Disease, Early Onset; Lewy Body Disease; Frontotemporal Lobar Degeneration
MeSH Terms: conditions — Alzheimer Disease; Lewy Body Disease; Frontotemporal Lobar Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to determine factors related to diagnosis delay for patients with young onset dementia (first symptoms before 60 years old) who live in North of France.

ELIGIBILITY:
Inclusion Criteria:

As part of this study, patients will be considered:

* Residing in the departments of Nord (59) and Pas-de-Calais (62),
* whose diagnosis of Alzheimer's disease or related illness (DLFT, DCL) was made and announced,
* Whose diagnosis of illness was made after 2007
* whose first symptoms appeared before the age of 60 Patients included in the COMAJ cohort and those who completed the Pathways medical and social booklet will have to meet these criteria to be selected for this study.

As part of the survey, caregivers of patients meeting the above criteria and the following two will be recruited:

* Having consulted or being followed by liberal neurologists or in hospital memory consultations (excluding CMRR-CNR-MAJ Lille) of the departments of Nord and Pas-de-Calais,
* Not monitored at the CMRR-CNR-MAJ Lille (ad hoc notice possible). The caregiver is defined as a family member or friend who helps regularly by doing the necessary tasks so that the sick person can keep as much autonomy as possible.

Exclusion Criteria:

* aged under 18
* no social coverage
* refusal to sign informed consent form

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of Alzheimer disease, Lewy Bodies Dementia or FrontoTemporal Lobar Degeneration and their caregivers
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
the delay between the diagnosis and the first symptomsIdentification of factors related with diagnosis delay | 10 years
  To determine the factors associated with diagnostic delay in young patients (early symptoms before age 60) with Alzheimer's disease or related degenerative disease (Fronto-temporal Lobar Degeneration , Lewy Body Dementia )

SECONDARY OUTCOMES:
Comparison of patient profiles followed at the CMRR-CNR-MAJ Lille and those who are not. | 10 years
  The different profiles are defined according to composite measures of socio-demographic type
Comparison of patients characteristics followed at the CMRR-CNR-MAJ Lille and those who are not.Impact of the diagnosis on YOD | 10 years
  The different characteristics are defined according to composite measures of socio-demographic type
the percentage of patients who have had a lack of information about the disease and possible aids | 10 years
  Identification of medico-social issues taht have been encountered by YOD patients during the care
the percentage of refusal or delay of treatment of certain medico-social aids by the competent authorities | 10 years
  Identification of medico-social issues taht have been encountered by YOD patients during the care

CONTACTS AND LOCATIONS:
Overall Officials: Florence Pasquier, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHRU, Lille, France